CLINICAL TRIAL: NCT00823576
Title: Efficacy of Ropivacaine Continuous Wound Instillation Versus Single Shot After Spine Fusion Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-CIR-03
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2022-11-29 (Actual); Status verified 2009-01

CONDITIONS: Postoperative Pain
Keywords: Arthodeses rachis lombar; Spinal Surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Group witness: one receiving a single bolus of analgesic
  Seepage simple person the end of intervention of 200mg of ropivacaïne 0,5 % at the level of zones it
  Interventions: Drug: Ropivacaine
- 2 (Active Comparator): Group catheter: receiving a single bolus of analgesic and an infiltration of Ropivacaine during 48 hours.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Compare the evolution of the postoperative levels of pain until J2, in the scheduled lumbar surgery between 2 groups of patients, one receiving a single bolus of analgesic, one receiving a single bolus of analgesic and an infiltration of Ropivacaine during 48 hours.

SUMMARY:
Because local anesthetic infiltration has not been comparated to continuous infusion after spine fusion surgery, the investigators designed this study to determine whether this technique could enhance analgesia and improve patient outcome after posterior lumbar arthrodesis.

The Main Objective of the study is to compare the evolution of the postoperative levels of pain until J2, in the scheduled lumbar surgery between 2 groups of patients, one receiving an infiltration "single shot" of local analgesic (Ropivacaïne), one receiving a single shot infiltration and a continuous infiltration of Ropivacaine during 48 hours.

In both groups the wound was infiltrated with a solution of ropivacaine 0.5% 200 mg/40 mL, and in one group an infusion of ropivacaine 0.2% 5 mL/h was maintained for 48 h.

The secondary outcomes are the consumption of morphine,the rate of the nausea and the postoperative vomits, the delay up to the first rise, the quality of the sleep, the duration of hospital stay and the persistence of residual pain.

DETAILED DESCRIPTION:
Postoperative pain after posterior lumbar stabilization surgery is related to soft tissue and muscle dissection and to manipulations and removal at the operation site. Most patients complain of severe pain at rest during the first 24 h after surgery. This pain increases considerably with mobilization because of the reflex spasm of paraspinal muscles that is triggered by the primary wound pain. During the following 48-72 h, postoperative back pain is generally moderate at rest, whereas it remains severe on movement and produces discomfort that can interfere with patient mobilization and, possibly, with discharge time. Despite the favourable effects of analgesia in the early postoperative period, this drug association may produce a number of well-known side effects, such as nausea, vomiting, respiratory depression, sedation, renal abnormality, and upper gastrointestinal and operative site bleeding. Local anesthetic infiltration of the surgical wound is a useful method in the treatment of postoperative pain after various surgical procedures. Ropivacaine is an interesting molecule for infiltration because of its vasoconstrictive properties and decreased neuro- and cardiotoxicity compared with bupivacaine.

The Main Objective of the study is to compare the evolution of the postoperative levels of pain until J2, in the scheduled lumbar surgery between 2 groups of patients, one receiving an infiltration "single shot" of local analgesic (Ropivacaïne), one receiving a single shot infiltration and a continuous infiltration of Ropivacaine during 48 hours.

After we obtained approval from the ethics committee and informed, written consent from patients, patients older than 18 years old , heavier than 50 kg, without psychological disorders, benefiting from of arthrodesis scheduled by a rachis lumbar posterior way were enrolled.

Patients were randomized to one of the two following postoperative analgesia groups after a presealed envelope was opened.

Post operative pain management is standardised with paracetamol, profenid and ACP morphine for each patient.

In both groups the wound was infiltrated with a solution of ropivacaine 0.5% 200 mg/40 mL, and in one group an infusion of ropivacaine 0.2% 5 mL/h was maintained for 48 h.

The Main Objective of the study is to compare the pain between 2 groups by means of the EVA (score of 0 for absence of pain in 10 for conceivable maximal pain) measured at H2, H8, H16, H24, H48.

The secondary outcomes are:

* The consumption of morphine 24 H and 48 H after surgery - The rate of the nausea and the postoperative vomits defined as the number of patients presenting the symptom on the number of patients in the group. - Delay up to the first rise
* Delay will be estimated in hours enter the end of the intervention surgery and the first one night
* The quality of the sleep estimated every morning with an analogical visual scale from 0 (very bad quality of sleep) to 10 (excellent quality of sleep)
* The duration of stay: calculated in days as the delay between the end of the intervention and the capacity at the exit.
* Recall of the patients in 3 and 6 months after the surgery to estimate the persistence of residual pains and if they still consume opioid. We shall ask to the patient to clarify the presence or the absence of pain The amount of analgesics required and the local and systemic adverse events were recorded for each patient.

Discharge was decided by the surgeons according to the following discharge criteria:1) satisfactory pain control for self-mobility; 2) uncomplicated wound-healing process 3) no impairments in haemoglobin 4) normothermie 5) normal transit, no nausea and vomit.

Sample-size calculation was based on an expected difference of 20 mm in VAS measurements for pain between groups. We calculate we need 64 patients for our main outcome. Each patient will be monitored during 6 month after the surgery.

The length of the study is 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients benefiting from of arthrodesis scheduled by a rachis lumbar posterior way
* Older than 18 years old
* Heavier than 50 kg
* Patients in the state health scheme
* Patients having signed consent

Exclusion Criteria:

* Surgery linked to an infectious, tumoral or traumatological cause
* Patients suffering of chronic pain define as patients consuming stage 3 analgesic since more than 3 months.- Patients receiving isoptine or flécaïne before surgery
* Arthrodesis on more than 3 stages
* Impossibility of cooperate with the patient
* Contra-indication for the maintain or the installation of a catheter diffusing analgesic
* Contra-indication of using local analgesic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-12; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Primary end points Principal: We compare the pain between 2 groups by means of the EVA (score of 0 for absence of pain in 10 for conceivable maximal pain) measured at H2, H8, H16, H24, H48. | 2 days

SECONDARY OUTCOMES:
The consumption of morphine mg-The rate of the nausea and the postoperative vomits defined-Delay up to the first rise-Delay will be estimated in hours enter the end of the intervention surgery and the first one night | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: LITRICO LS Stéphane, PH, Principal Investigator — CHU de Nice - Hôpital Pasteur - 30 ave de la Voie Romaine - 06100 Nice
Locations (1):
- CHU de Nice - 4 avenue Reine Victoria - Hôpital de Cimiez, Nice, Alpes-Maritimes, France